CLINICAL TRIAL: NCT02674906
Title: Exposure of Salvaged Blood to Inflammation and Oxidative Stress: the Effect of Different Anticoagulant Regimes. Heparin vs Citrate in Cellsaver (HECICS).
Brief Title: Exposure of Salvaged Blood to Inflammation and Oxidative Stress: the Effect of Different Anticoagulant Regimes (HECICS)
Acronym: HECICS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ziekenhuis Oost-Limburg (Other)
Responsible Party: Principal Investigator, Willem Boer, Consultant Intensivist, Ziekenhuis Oost-Limburg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: HECICS
Record Dates: First submitted 2016-01-24; First posted 2016-02-05 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Intra Operative Bleeding, Blood Salvage
MeSH Terms: interventions — Heparin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- citrate (Active Comparator): A quantity of 20 ml ACD-A per 100 ml of collected blood is used to prevent coagulation in the cell savage process. Pre-prepared ACD-A solutions is available (composition of ACD-A solution used: 22.0 g sodium citrate dehydrate, 24.5 g glucose monohydrate, 8.0 g citric acid monohydrate per 1000 ml of water
  Interventions: Drug: ACD-A
- heparin (Active Comparator): A heparinised saline solution of 25,000 IU of heparin per 1 litre of intravenous normal saline (0.9% NaCl) solution is used with a dosage of 20 ml of solution per 100 ml of collected blood. This type of solution is not commercially available and is made locally. This solution is used in the cell salvage process to prevent coagulation.
  Interventions: Drug: Heparin

INTERVENTIONS:
Drug: ACD-A — use of ACD-A as anticoagulant after blood salvage during cardiac surgery
  Other Names: Anticoagulant Citrate Dextrose Solution--Formula A
  Arms: citrate
Drug: Heparin — use of heparin as anticoagulant after blood salvage during cardiac surgery
  Other Names: heparin sodium
  Arms: heparin

SUMMARY:
The primary aim of this randomized controlled study is to determine whether the use Anticoagulant Citrate Dextrose Solution--Formula A (ACD-A) in cell salvage reduces inflammation and oxidative stress in cell saver blood compared to heparin. The secondary aim is to determine whether any differences in activation can be correlated to any differences in postoperative clinical outcome.

DETAILED DESCRIPTION:
The first primary outcome of this study is the difference in concentration of pro- and anti-inflammatory markers and markers of oxidative stress in the cell-free fraction of the centrifugate of the unwashed autologous blood/anticoagulant mixture in the cell saver reservoir, after correction for cardiopulmonary bypass (CPB) time up to the start of the first washing cycle and contact time of the anticoagulant (either ACD A or heparin) with the saved blood:

* total antioxidant status (TAS)
* Total thiols in proteins (TTP)
* oxidized LDL (oxLDL)
* Pro-inflammatory markers: interleukins (IL), IL-6, IL-8, myeloperoxidase (MPO)
* Anti-inflammatory marker: IL-10

The second primary outcome of this study is the difference in direct quality of the washed, salvaged red blood cells (RBC):

* Blood smear: evaluation by light microscopy
* Osmotic fragility
* Haemoglobin and hematocrit
* Free haemoglobin
* Free iron
* Lactate
* pH Confounding factors (CPB duration, contact time of anticoagulant with saved blood, time since first washing cycle in case of multiple washing cycles) will be controlled for.

Secondary outcome:

The difference in concentration of the same pro/anti-inflammatory and oxidative stress markers in patient plasma preoperatively vs immediately before and after transfusion of cell saver blood (2 to 3 hours after transfusion and before extubation or transfusion of allogenous blood).

* C-reactive protein (CRP)
* TAS, TTP
* oxLDL
* IL-6, IL-8, IL-10
* MPO Markers for hemolysis in patient plasma preoperatively vs immediately pre- and post-transfusion of the salvaged RBC (indirect quality of the washed salvaged RBC).
* Free Hb
* Free iron, ferritin, transferrin
* Haptoglobin
* Hepcidin

ELIGIBILITY:
Inclusion Criteria:

Elective cardiac revascularization surgery patients: subgroup analysis for

* on pump coronary artery bypass grafting (CABG)
* off pump CABG (OPCABG)

Exclusion Criteria:

* Urgent procedures
* Severe shock
* Active infection
* Inflammatory diseases
* Active neoplasia
* Immune suppressive drugs
* Active or recent renal replacement therapy (RRT)
* Anticoagulation or anti-aggregation therapy that hasn't been timely interrupted according to guidelines (12,13)
* Need for allogenous blood transfusion before completion of data collection
* Massive peroperative bleeding that cannot be safely managed while collecting study data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
difference in concentration of pro- and anti-inflammatory markers and markers of oxidative stress in the cell-free fraction of the centrifugate of the unwashed autologous blood/anticoagulant mixture in the cell saver reservoir | maximum 3 hours post-operatively
  measurement of: TAS: total antioxidant status TTP: total thiols in proteins oxLDL: oxidized LDL Pro-inflammatory markers: IL-6, IL-8, myeloperoxidase (MPO) Anti-inflammatory marker: IL-10

SECONDARY OUTCOMES:
The second primary outcome of this study is the difference in direct quality of the washed, salvaged RBC: | maximum 3 hours post-operatively
  The second primary outcome of this study is the difference in direct quality of the washed, salvaged RBC:
  Blood smear: evaluation by light microscopy Osmotic fragility Haemoglobin and hematocrit Free haemoglobin Free iron Lactate pH

CONTACTS AND LOCATIONS:
Locations (1):
- Ziekenhuis Oost-Limburg, Genk, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Boer W, van Tornout M, Brusseleers M, Strauven M, de Vooght P, Vander Laenen M, Hoste E, Jorens PG. The effects of differing anticoagulant regimes on blood quality after cell salvage in coronary artery bypass grafting (CABG): a pilot study. J Cardiothorac Surg. 2023 Apr 8;18(1):116. doi: 10.1186/s13019-023-02246-w. PMID 37031168